CLINICAL TRIAL: NCT00161967
Title: Open-label Follow-up Study to Investigate the Seropersistence of TBE Antibodies and the Booster Response to a Tick-borne Encephalitis Vaccine in Children and Adolescents Aged 3 - 18 Years
Brief Title: TBE Antibody Persistence and Booster Vaccination Study in Children and Adolescents (Follow-up to Study 209)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Martin Kraft, Clinical Project Manager, Baxter Healthcare Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 700401
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-Borne
Keywords: tick-borne encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated) — Subjects receive one vaccination with either FSME-IMMUN 0.25 ml or FSME-IMMUN 0.5 ml, depending on their age.

SUMMARY:
The purpose of this study is to assess the seropersistence of TBE antibodies in children and adolescents aged 1 to 15 years at the time of their first vaccination, 24 months and 34 months after completion of primary immunization with FSME-IMMUN 0.25 ml (3 vaccinations during the predecessor study 209), as well as the immune response to a booster vaccination with FSME-IMMUN 0.25 ml or FSME-IMMUN 0.5 ml administered 36 months after the third vaccination (in Study 209).

Protocol amendment of October 2006: The study has been prolonged for children and adolescents who still showed highly positive TBE virus antibody concentrations at approximately 3 years after the third vaccination and therefore did not receive a booster vaccination at this time point. Further follow-up of TBE antibody persistence is now included for these subjects at 46 and 58 months after the third vaccination (in Study 209), as well as a booster vaccination offered at either 48 or 60 months after the third vaccination (in Study 209), depending on individual TBE antibody levels.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Baxter study 209 and:
* They and/or their parents / legal guardians understand the nature of the study and agree to its provisions
* Written informed consent is available from the parents / legal guardians according to national law
* Written informed assent is available from the child/adolescent according to age and capacity of understanding
* They received the third vaccination with FSME-IMMUN 0.25 ml during the course of Baxter study 209
* Blood was drawn after their third vaccination during the course of Baxter study 209
* They showed an ELISA concentration > 126 VIE U/ml and / or a NT titer >=10 after the third vaccination in Baxter study 209
* They or their parents / legal guardians agree to keep a Subject Diary

Exclusion Criteria:

* Received any TBE vaccination since their third vaccination with FSME-IMMUN 0.25 ml
* Have a history of infection with or vaccination against other flaviviruses (Dengue fever, yellow fever and / or Japanese B-encephalitis virus) since their third vaccination with FSME-IMMUN 0.25 ml
* Are known to be HIV positive (a special HIV test is not required for the purpose of the study) since their third vaccination with FSME-IMMUN 0.25 ml
* Received a blood transfusion or immunoglobulins within 30 days of the first and second blood draw (as applicable)
* Have a known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent level of other alcoholic beverages)
* Have participated in another Baxter vaccine study within the last six months (with the exception of follow-up studies)

Subjects will not be eligible for booster vaccination if they:

* Do not meet the inclusion / exclusion criteria
* Are not clinically healthy, (i.e. the physician would have reservations vaccinating with a TBE vaccine outside the scope of a clinical trial)
* Suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions
* Have shown an allergic reaction to one of the components of the vaccine since their third vaccination in Baxter study 209
* Have donated blood or plasma within 30 days of the booster vaccination if female of childbearing potential - are pregnant or breastfeeding before the booster vaccination (positive pregnancy test result at the medical examination before the booster vaccination)
* Are simultaneously participating in another clinical trial including administration of an investigational product within six weeks prior to the booster vaccination until the end of the study

Subjects who meet the inclusion/exclusion criteria, but have a febrile illness (body temperature >=38.0°C, measured orally) at the scheduled time of vaccination will not be vaccinated until their body temperature returns to normal.

Subjects who received any vaccination within 4 weeks prior to the booster vaccination will not be vaccinated until an interval of four weeks has passed.

If subjects received antipyretics within 4 hours prior to the intended TBE vaccination, the vaccination should be performed at a later time.

Females of childbearing potential will only be vaccinated if they agree to employ adequate birth control measures from 4 weeks before the booster vaccination until the end of the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 375 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Seropositivity rate measured by ELISA and/or NT according to Adner et al., 2001 at each available time point after the third vaccination in study 209 and separately at each available time point after the booster vaccination in this study | TBE virus antibody tests at pre-determined intervals with the last test at 21-35 days after the booster vaccination in this study

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter BioScience
Locations (3):
- Grieskirchner Strasse 17, Wels, Upper Austria, Austria
- Hauptstrasse 240, Kehl, Germany
- Niepubliczny ZOZ, Zamość, Poland